CLINICAL TRIAL: NCT01019603
Title: A Single-Center, Randomized, Open-Label Study to Evaluate the Bioavailability of Tazarotene Foam, 0.1%, and Tazorac Gel, 0.1%, in Subjects With Acne Vulgaris
Brief Title: A Study to Evaluate the Bioavailability of Tazarotene Foam, 0.1%, and Tazorac Gel, 0.1%, in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 114565
Record Dates: First submitted 2009-11-19; First posted 2009-11-25 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — tazarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tazarotene foam 0.1%
  Interventions: Drug: Tazarotene
- 2 (Active Comparator): Tazaroc Gel 0.1%
  Interventions: Drug: Tazaroc Gel

INTERVENTIONS:
Drug: Tazarotene — Topical Tazarotene foam applied daily for 22 days.
  Other Names: Tazorac
  Arms: 1
Drug: Tazaroc Gel — Topical tazarotene gel applied daily for 22 days.
  Other Names: Tazorac
  Arms: 2

SUMMARY:
The purpose of this study is to assess systemic exposure of a new foam formulation of tazarotene, 0.1% compared with Tazorac Gel, 0.1%. The study design and dosing regimen are based on previous clinical studies with Tazorac Gel and Tazorac Cream.

DETAILED DESCRIPTION:
A single-center, randomized, open-label, phase 1, comparative bioavailability study in subjects with moderate to severe acne vulgaris. Approximately 30 subjects will be enrolled and randomized to 1 of the 2 study product groups in a 1:1 ratio (tazarotene foam: Tazorac Gel). Study product will be applied once daily for 22 days to the face, upper chest, upper back, and shoulders. Following the baseline visit, subjects will return to the study center daily for study product application. Blood samples to determine plasma concentrations of tazarotenic acid will be collected before study product application on days 1, 8, 12, 15, 18, 20, and 22, and collected at multiple time points over a 72 hour period on days 22 through 25.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 12 years of age or older who is in good general health.
* Have an Investigator's Static Global Assessment (ISGA) score of 3 or greater at baseline. The area considered for the ISGA must be confined to the face.
* Regular menstrual cycle prior to study entry (as reported by the subject) for females of childbearing potential.
* Negative urine pregnancy test for females of childbearing potential. • Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses.

Women who are not currently sexually active must agree to use medically accepted methods of contraception should they become sexually active while participating in the study. Male subjects and/or their partners must use a medically acceptable form of contraception.

* Nonsmoker or smoker with at least 30 days abstinence from smoking or using nicotine-containing products prior to study entry and willing not to smoke or to use nicotine-containing products throughout the study.
* Ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study.
* Capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol specific procedures are performed

Exclusion Criteria:

* Female who is pregnant, trying to become pregnant, or breast feeding.
* History of known or suspected intolerance to any of the ingredients of the study products.
* Use of topical antibiotics or topical corticosteroids for acne treatment within the past 2 weeks.
* Use of systemic corticosteroids within the past 4 weeks.
* Use of systemic retinoids (eg, isotretinoin) within the past 6 months.
* Concurrent use of medications known to be photosensitizers because of the possibility of augmented photosensitivity.
* Use of topical anti-acne medications (eg, benzoyl peroxide, retinoids) within the past 2 weeks.
* Concomitant use of of facial products such as: abradants, facials, peels containing glycolic or other acids .
* Facial procedure (eg, chemical or laser peel or microdermabrasion) performed by an esthetician, beautician, physician, nurse, or other practitioner within the past 2 weeks.
* History or evidence of skin conditions other than acne (eg, eczema) that would interfere with the subject's participation in the study.
* Consumption of alcohol within 24 hours prior to study product application on days 8, 12, 15, 18, 20, and 22 and within 72 hours post application on day 22.
* Consumption of xanthine-containing beverages or products (eg, caffeinated coffee, tea, over-the counter medication for cold symptoms) within 24 hours prior to study product application on days 8, 12, 15, 18, 20, and 22 and within 72 hours post-application on day 22.
* Anticipated need to engage in activities or exercise that would cause profuse sweating during the study.
* Anticipated need for surgery or hospitalization during the study.
* Require or desire excessive or prolonged exposure to ultraviolet light (eg, sunlight or tanning beds) during the study.
* Concurrent involvement in another investigational study or participation within 30 days prior to the start of this study.
* Any other condition that, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.
* Currently lives in the same household as currently enrolled subjects; is an employee of Stiefel, an investigator, or a contract research organization involved in the study; or is an immediate family member (eg, partner, offspring, parents) of an employee involved in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10-12 (Actual); Primary Completion 2009-12-20 (Actual); Study Completion 2009-12-20 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of tazarotenic acid in subjects with acne vulgaris | Days 1, 8, 12, 15, 18, 20, 22 (pre-dose and 3, 4.5, 6, 7.5, 9, 12, 16, 20, 24, 38, 48, 62, and 72 hr post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- DermResearch, Inc., Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Jarratt M, Werner CP, Alio Saenz AB. Tazarotene foam versus tazarotene gel: a randomized relative bioavailability study in acne vulgaris. Clin Drug Investig. 2013 Apr;33(4):283-9. doi: 10.1007/s40261-013-0065-1. PMID 23456673
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114565 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114565?search=study&search_terms=114565#rs
- Available data/document: Statistical Analysis Plan: 114565 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114565 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114565 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114565 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114565 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114565 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114565 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register